CLINICAL TRIAL: NCT05598645
Title: Thulium Fiber Laser (TFL) Versus Holmium MOSES Laser in Ureteroscopic Management of Kidney Stones 10-20mm: A Randomized Prospective Clinical Trial
Brief Title: Thulium Fiber Laser (TFL) Versus Holmium MOSES Laser for Ureteroscopic Management of Kidney Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-791
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thulium Fibre Laser (TFL) (Experimental): Patients randomized to this arm will undergo treatment using the TFL.
  Interventions: Device: Thulium Fibre Laser
- MOSES Holmium Laser (Experimental): Patients randomized to this arm will undergo treatment using the MOSES Holmium laser.
  Interventions: Device: MOSES Holmium Laser

INTERVENTIONS:
Device: Thulium Fibre Laser — Participants will undergo treatment using the TFL
  Arms: Thulium Fibre Laser (TFL)
Device: MOSES Holmium Laser — Participants will undergo treatment using the MOSES Holmium laser.
  Arms: MOSES Holmium Laser

SUMMARY:
This study aims to compare the efficacy and safety of both types of lasers, Holmium MOSES and TFL, in management of kidney stones requiring treatment.

DETAILED DESCRIPTION:
The prevalence of kidney stones has been increasing over the last two decades with lifetime recurrence risk reported to be as high as 50%. Holmium lasers are nowadays considered the "gold standard" for treatment of urinary tract stones.

Recently, the holmium laser urology platform from Lumenis has been updated to include a new technology called MOSES, which provides improved energy delivery of the laser to treat the stones, reduces migration of the stone during the procedure, and limits potential collateral tissue damage.

A new generation of lasers has evolved due to the advances in laser fiber technology, leading to the development of the Thulium Fiber Laser (TFL). TFL can operate within a large range of energy, frequency and pulse duration settings. The small fiber size is one of the main advantages of TFL, as it allows better endoscope performance through easier deflection and bigger working channel space. Furthermore, it produces small stone fragments and better dusting capabilities compared to the standard Holmium laser when adjusted on the same power settings.

This study will compare the efficacy and safety of Holmium MOSES and TFL in management of kidney stones requiring treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and over at the time of enrollment.
2. Patients referred with single kidney stones of 10-20 mm in its largest diameter, or multiple stones involving a single calyx.
3. Written informed consent to participate in the study
4. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

1. Patients with ipsilateral distal ureteral stones or stricture.
2. Stone size > 20 mm or multiple kidney stones in different calyces.
3. Previous shock wave lithotripsy (SWL) treatment for the same stone.
4. Participants with active urinary tract infection until appropriately treated
5. Uncorrected coagulopathy (anticoagulants or blood thinners which cannot be withheld before surgery).
6. Pregnancy.
7. Participants with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study.
8. Participants who are uncooperative or cannot follow instructions.
9. Participants who lack the capacity, or cannot speak English, in order to provide free and informed written consent.
10. Patients with solitary kidney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Procedural Time | Intraoperative
  Measured in number of minutes from the insertion of the ureteroscope to the removal of the ureteroscope.

SECONDARY OUTCOMES:
Stone Free Rate (SFR) | 4 and 12 weeks post-op
  SRF will be defined as the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the urinary tract which were defined as ˂4 mm, asymptomatic, non-obstructive and non-infectious stone particles.
Total operative time | Intraoperative
  Measured in n minutes from the anesthesia induction until placement of the stent.
Lasing time | Intraoperative
  Measured in minutes and defined as the time the laser was in use, not including pedal pauses.
Total energy used | Intraoperative
  Measured in kilojoules, defined as energy used to fragment the stones into small pieces (≤2 mm).
Laser efficiency | Intraoperative
  Measured as mm per minute and defined as the stone size (mm) that can be treated every minute; the cumulative stone size (adding the maximum size of each stone that is treated during the surgery) is divided by the lasering time.
Number of times the laser pedals are pressed | Intraoperative
  Measured as a numerical value, defined as number of left, right, and total pedal presses
Percentage of Patients with Post-op Complications | 4 weeks
  Percentage of patients that results with a post-op complication

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Elmansy, MD, Principal Investigator — Urologist
Locations (1):
- Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No